CLINICAL TRIAL: NCT01401205
Title: The Predictor of Respiratory Discomfort After the Shoulder Arthroscopic Surgery as Measured by Upper Airway Ultrasonography
Brief Title: The Predictor of Respiratory Discomfort After the Shoulder Arthroscopic Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sujoo Choi, Professor, Samsung Medical Center
Other Study IDs: 2011-06-028
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Shoulder Arthroscopic Surgery
Keywords: shoulder arthroscopic surgery; dyspnea; airway diameter
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- shoulder arthroscopic surgery group: the patients who undergo the elective shoulder arthroscopic surgery of rotator cuff repair
  Interventions: Other: upper airway ultrasonographic examination

INTERVENTIONS:
Other: upper airway ultrasonographic examination — upper airway ultrasonographic examination and cuff leak test
  Other Names: upper airway ultrasonographic examination ,; cuff leak test

SUMMARY:
The investigators applied upper airway ultrasonographic examination focusing the measurement of upper airway diameters in patients undergoing shoulder arthroscopic surgery to evaluate the change of upper airway anatomy before and after the surgery. The investigators also tried to find any findings of ultrasonographic examination that could reliably predict the dyspnea or airway compression after extubation. The investigators tried to compare the ultrasonographic findings with those of chest radiograph to validate the measurements of the ultrasonographic examination. A cuff leak test was preformed to evaluate its ability to predict the upper airway obstruction in shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
During shoulder arthroscopic surgery, extravasation of irrigation fluid can occur around the shoulder and trachea, compressing the upper airway. Although the extravasation is generally reabsorbed asymptomatically within 12 hours, there are cases that lead to reintubation or life-threatening complications.

An endotracheal tube is the most reliable method of securing the airway from airway obstruction during a shoulder arthroscopy surgery. However, since the airway may become obstructed after extubation, airway patency should be verified before extubation. Direct visualization of the larynx or trachea using laryngoscopy or bronchoscopy is difficult due to the presence of the tracheal tube. A cuff leak around the tracheal tube in a cuff-deflated condition is suggested to be a predictor of successful extubation. However, its reliability has been questioned in adult patients. A cuff leak could be affected by paratracheal pressure, which is thought to be elevated during shoulder arthroscopy. In a recent study, it was shown that laryngeal ultrasound can be a reliable, non-invasive method for the evaluation of laryngeal morphology or predicting post-extubation stridor.

The investigators applied upper airway ultrasonographic examination focusing the measurement of upper airway diameters in patients undergoing shoulder arthroscopic surgery to evaluate the change of upper airway anatomy before and after the surgery. The investigators also tried to find any findings of ultrasonographic examination that could reliably predict the dyspnea or airway compression after extubation. The investigators tried to compare the ultrasonographic findings with those of chest radiograph to validate the measurements of the ultrasonographic examination. A cuff leak test was preformed to evaluate its ability to predict the upper airway obstruction in shoulder arthroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective shoulder arthroscopic surgery (rotator cuff repair)

Exclusion Criteria:

* patients with airway anomaly
* patients with anticipated difficult airway
* patients with hemodynamic unstability
* patients with severe cardiopulmonary disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective shoulder arthroscopic surgery (rotator cuff repair)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Airway transverse diameter | 10 min before anesthesia induction
  airway transverses diameter measured on the upper airway ultrasonographic image: measure at three level (vocal cord, subglottis, trachea)
Airway transverse diameter | 20 min after end of surgery
  airway transverses diameter measured on the upper airway ultrasonographic image: measure at three level (vocal cord, subglottis, trachea)

SECONDARY OUTCOMES:
depth of skin to airway anterior border | 10 min before anesthesia induction and 20 min after the surgery
  depth of skin to airway anterior border measured at three levels: vocal cord, subglottis, trachea level
depth of skin to pleura | 10 min before anesthesia induction and 20 min after the end of surgery
  bilateral depth of skin to pleura at first and third intercostal space on the midclavicualr line measuread on the ultrasonographic image
endotracheal tube balloon cuff pressure | 10 min after anesthesia induction and 60 min after surgery start
  endotracheal tube balloon cuff pressure
percent cuff leak | 10 min after anesthesia induction and 60 min after surgery start
  The difference in the actual exhaled volume between the averages of pre- and post-cuff deflation was calculated. This number was divided by the tidal volume before cuff deflation and multiplied by 100. The resulting number was recorded as the percent cuff leak.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Joo Choi, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea